CLINICAL TRIAL: NCT01134991
Title: Pilot, Randomized, Double Blind, Placebo Controlled, Parallel Group, Dose Range Finding Study, to Evaluate the Tolerability and Safety of FXFM244 Antibiotic Foam and to Monitor Its Clinical Effect in Moderate to Severe Rosacea Patients
Brief Title: Study to Evaluate the Safety and Efficacy of Topical Minocycline FXFM244 in Rosacea Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0041-10LND /FX2010-02
Record Dates: First submitted 2010-05-26; First posted 2010-06-02 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2010-08

CONDITIONS: Rosacea
Keywords: rosacea; topical; minocycline; foam; phase II
MeSH Terms: conditions — Rosacea; cyclopia sequence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Topical Minocycline Foam FXFM244 Placebo (Placebo Comparator): Minocycline Foam FXFM244 Placebo
  Interventions: Drug: Topical Minocycline Foam FXFM244
- Topical Minocycline Foam FXFM244, 1% (Experimental): Minocycline Foam FXFM244, 1%
  Interventions: Drug: Topical Minocycline Foam FXFM244
- Topical Minocycline Foam FXFM244, 4% (Experimental): Minocycline Foam FXFM244, 4%
  Interventions: Drug: Topical Minocycline Foam FXFM244

INTERVENTIONS:
Drug: Topical Minocycline Foam FXFM244 — FXFM244 - 1%, FXFM244 - 4% or Placebo to be applied twice daily during 12 weeks

SUMMARY:
Acne rosacea is a chronic acneiform disorder affecting both the skin and the eye. It is a syndrome of undetermined etiology characterized by both vascular and papulopustular components involving the face and occasionally the neck and upper trunk.

This is a pilot phase II study to evaluate the tolerability and safety and to monitor the clinical efficacy of Topical Minocycline Foam FXFM244 in moderate to severe Rosacea patients.

DETAILED DESCRIPTION:
A Pilot, Randomized, Double Blind, Placebo Controlled, Parallel Group, Dose Range Finding Study. The study will involve three treatment groups. Eligible patients will be randomized to receive either FXFM244 - 1%, FXFM244 - 4% or Placebo, in a blinded fashion. Patients will be treated twice daily for 12 weeks. Following the screening period and baseline visit, study subjects will return at Weeks 3, 6, 9 and 12. A follow up visit will take place at week 16. At each visit, patients will be evaluated via lesion count, global assessment tolerability and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical diagnosis of moderate to severe facial rosacea as determined by:

   * At least 8 but no more than 50 total papules and/or pustules (inflammatory lesions)
   * Presence of moderate to severe erythema
   * Presence of telangiectasia.
   * An Overall Rosacea Severity score ≥2.5
2. Patient is male or female over 18 years of age.
3. No known medical conditions that, in the Investigator's opinion could interfere with study participation
4. Patient is willing and able to comply with all requirement of the protocol
5. Patient is willing and able to give written informed consent prior to participation in the study

Exclusion Criteria:

1. Presence of skin diseases at or near the investigational area
2. Immunosuppressed state or other serious systemic disease
3. Signs and/or symptoms of systemic infection
4. Concomitant medication:

   * Use of oral and/or topical antibiotic treatment within 14 days prior to study entry.
   * Use of any topical anti-rosacea agent except antibiotics within 14 days prior to study entry.
   * Use of cyproterone acetate, CPA-containing contraceptives (e.g. Diane) or other corticosteroids (during the last 3 months);
   * Use of retinoids (during the last 4 weeks)
5. Use of artificial sun bath or having a sun holiday during the last 2 weeks
6. Alcohol or drug abuse, according to assessment by the investigator
7. Known or suspected hypersensitivity to Minocycline or any of the excipients in the Study Medication
8. Use of another investigational drug within 30 days prior to entry into this study
9. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-06; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Improvement in signs and symptoms of rosacea | 12 weeks

SECONDARY OUTCOMES:
The severity of the overall rosacea condition will be measured at baseline and at all follow-up visits. The severity will be assessed and graded based on the scales for erythema, telangiectases and number of papulopustular lesions | 0, 3, 6, 9 and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel